CLINICAL TRIAL: NCT02409212
Title: Exercise Training as a Novel Primary Therapy for Men With Localised Prostate Cancer: the PANTERA Trial (Prostate cAncer Novel ThERApy)
Brief Title: Exercise Training as a Novel Primary Therapy for Men With Localised Prostate Cancer
Acronym: PANTERA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other); University of Sheffield (Other); Queen Mary University of London (Other); University College London Hospitals (Other); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH 18624
Record Dates: First submitted 2015-01-20; First posted 2015-04-06 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): 12 months of aerobic exercise training with behaviour change support
  Interventions: Behavioral: Aerobic exercise training
- Comparison (Placebo Comparator): Optimal active surveillance according to NICE guidelines and written exercise guidelines from Macmillan cancer
  Interventions: Behavioral: Placebo surveillance and written exercise guidelines

INTERVENTIONS:
Behavioral: Aerobic exercise training — Aerobic exercise training will be undertaken for 12 months, combining supervised and independent exercise sessions. Behaviour change counselling will take place bi-monthly, either via face to face sessions during exercise or via telephone by study clinical exercise specialist according to participant preference.
  Arms: Intervention
Behavioral: Placebo surveillance and written exercise guidelines — Optimal active surveillance according to NICE guidelines and written exercise guidelines from Macmillan cancer
  Arms: Comparison

SUMMARY:
Study design: The study is a two arm randomised controlled trial (randomisation ratio 1:1) comparing an aerobic exercise training intervention to usual care plus exercise advice. The primary outcome is the feasibility of the intervention as novel primary therapy in men with localised prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

In accordance with NICE active surveillance guidelines, men:

* Who have been evaluated using a combination of clinical, bio-chemical, imaging and/or biopsy, within the last 12 months
* With histologically confirmed low or intermediate risk prostate cancer, Gleason score ≤7 (3+4, not 4+3)
* With up to T2a clinical stage tumours
* With pre-treatment PSA ≤20 ng/mL
* Who are willing to participate in optimal active surveillance and provide written informed consent
* With life expectancy of ≥10 years

Exclusion Criteria:

Men:

* With unstable angina
* With uncontrolled hypertension
* With recent myocardial infarction (within the past 6 months)
* With pacemakers
* Already undertaking regular physical activity (greater than 90 minutes of moderate intensity exercise, per week) will be excluded
* With any other physical or mental limitation preventing participation in trial assessments
* Participating in other clinical trials which might bias the evaluation of the primary objectives of the present study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by rate of recruitment | 36 months
  The rate of recruitment will be measured by comparing the number of patients screended to the number of patients recruited. This will allow us to asses if a future full-scale trial is feasible.

SECONDARY OUTCOMES:
Feasibility as measured by Intervention adherence | 36 months
  Intervention adherence will be assessed using an exercise log book and heart rate monitor to objectively record independent exercise behaviour and support adherence and compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Rosario, MD, Principal Investigator — University of Sheffield / Sheffield Teaching Hospitals
Locations (1):
- Sheffield Teaching Hospitals NHS Trust, Sheffield, South Yorkshire, United Kingdom